CLINICAL TRIAL: NCT05783778
Title: Evaluation of the Role of Latent Toxoplasmosis in Female Patients With Active Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zineb Gamee Aly Ahmed, Zienab Gamea Ali Ahmed, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-03-05MS
Record Dates: First submitted 2023-03-08; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Acne Vulgaris; Toxoplasmosis
MeSH Terms: conditions — Acne Vulgaris; Toxoplasmosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toxoplasmosis seropositive female patients with active acne vulgaris (Experimental)
  Interventions: Diagnostic Test: Free testosterone levels and toxoplasma igG
- Toxoplasmosis seronegative in female patients with active acne vulgaris (Experimental)
  Interventions: Diagnostic Test: Free testosterone levels and toxoplasma igG

INTERVENTIONS:
Diagnostic Test: Free testosterone levels and toxoplasma igG — Free testosterone levels and toxoplasma igG in serum by ELISA

SUMMARY:
Acne vulgaris is one if the most common chronic inflammatory skin disorders.Acne is characterized by forming of inflammatory and non inflammatory lesions mainly on the Face,neck,arms, upper trunk and back

DETAILED DESCRIPTION:
One of the hidden hormonal imbalance is Toxoplasma infection.Toxoplasmosis is a zoonotic infection the definite host is feline whereas human and other warm blooded animals are intermediate host . Endocrine alterations occuring during toxoplasmosis can be a hidden cause of acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

- Female patients with active acne vulgaris

Exclusion Criteria:

* Patients with history of hormonal treatment Patients received anti toxoplasma therapy Patients with dermatological diseases caused by hormonal disturbances Pregnant and lactating patients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Measuring Toxoplasma igG and free testosterone in acne vulgaris patients and controls | One month
  Detect if the toxoplasma latent infection can be associated with disease severity and hormonal disturbances in acne vulgaris female patients

IPD SHARING:
Plan to Share IPD: Undecided